CLINICAL TRIAL: NCT03225443
Title: Shanghai First Maternity and Infant Hospital
Brief Title: Observation and Evaluation of Short-term Curative Effect of Local Advanced Cervical Cancer Treated With Particle Radiotherapy Versus Neoadjuvant Chemotherapy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Shanghai First Maternity and Infant Hospital (Other)
Collaborators: RenJi Hospital (Other); Shanghai Proton and Heavy Ion Center (Other)
Responsible Party: Sponsor
Other Study IDs: Xiaoqing Guo
Record Dates: First submitted 2017-07-19; First posted 2017-07-21 (Actual); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Uterine Cervical Neoplasms; Locally Advanced Cervical Cancer
Keywords: Locally advanced cervical cancer; Particle radiotherapy; Neoadjuvant Chemotherapy
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Particle Radiotherapy: The patients will receive particle radiotherapy before operation,and then radical hysterectomy, removal of pelvic lymph nodes and abdominal aorta lymph nodes would be conducted. Besides ovary reservation would be made according to the individual situation. Concurrent radiation and chemotherapy would be performed according to the clinical situation.
- Neoadjuvant Chemotherapy: The patients will receive NACT before operation,and then radical hysterectomy, removal of pelvic lymph nodes and abdominal aorta lymph nodes would be conducted. Besides ovary reservation would be made according to the individual situation. Concurrent radiation and chemotherapy would be performed according to the clinical situation.

SUMMARY:
Locally advanced cervical cancer (LACC) refers to the clinically cervical visible lesion with a diameter of > 4 cm, which has been considered as a high risk of early cervical cancer for a long time. Because of local bulk lesion of LACC, the risk of radical hysterectomy is pretty high and the radical effect commonly does not meet the satisfactory. Therefore, 1-3 course of neoadjuvant chemotherapy (NACT) were carried out before operation. However, nearly 20% of patients are not sensitive to NACT. Therefore NACT did not bring any benefits to radical surgery even to some extent delayed the treatment.

Traditional radiotherapy is also commonly used in the treatment of LACC, however ovarian function would be permanently destroyed especially for young patients, additionally radioactive complications to adjacent organs of cervical such as vagina, bladder and rectal also commonly happened, moreover sexual dysfunction after radiotherapy significantly affect the life quality of young patients.

Particle radiotherapy developed recently, has the advantages of short course of treatment and mild side effects, due to its special working mechanism, Bragg effect. So the amount of radiation in the tumor tissue is very extremely high, and in the adjacent tissue is quiet low, therefore the organs at risk were protected by avoiding unnecessary damage.

Based on these, we proposed the application of particle radiotherapy in LACC pre-operation, and comprehensively evaluated recent curative effect, complications and long-term follow-up between particle radiotherapy and NACT. Furthermore, the clinical significance and long-term application prospects about particle therapy were objectively assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Pathological diagnosis: squamous carcinoma, adenocarcinoma, adenosquamous carcinoma
2. The pathological staging: IB2，IIA2

Exclusion Criteria:

Underwent surgery or radiation and chemotherapy

Sex: Female
Age Groups: Child, Adult, Older Adult
Study Population: All patients from Sep 2017 until Sep 2020 in Shanghai First Maternity and Infant Hospital, Tongji University and Renji Hospital Shanghai Jiaotong University School of Medicine.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2017-09-30 (Estimated); Primary Completion 2020-09-30 (Estimated); Study Completion 2020-09-30 (Estimated)

PRIMARY OUTCOMES:
The recurrence rate | 3 years after treatment

SECONDARY OUTCOMES:
The transfer rate | 3 years after treatment
mortality | 3 years after treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai First Maternity and Infant Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided